CLINICAL TRIAL: NCT01948934
Title: Clinic Trial in Phase 1 Using Amniotic Membrane for the Skin Replacement in Big Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA/GH; 2011-004395-11 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Wound
Keywords: Skin; Injury; Membrane amniotic; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- amniotic membrane in big wounds (Experimental): The wound will be washed with saline and debrided if necessary. Control microbiological cultures will be taken and applied amniotic membrane fragments sufficient to cover the wound, putting in contact the basement membrane of the AM with granulation tissue
  Interventions: Procedure: Amniotic membrane in big wounds

INTERVENTIONS:
Procedure: Amniotic membrane in big wounds — The wound will be washed with saline and debrided if necessary. Control microbiological cultures will be taken and applied amniotic membrane fragments sufficient to cover the wound, putting in contact the basement membrane of the AM with granulation tissue

SUMMARY:
The purpose of this study is to determine the safety of use of a new therapeutic strategy for the treatment of patients with large wounds

DETAILED DESCRIPTION:
Amniotic membrane (AM) is a useful tissue as a biological dressing with numerous advantages it has a very similar structure to the skin and his biological and immunological properties.

ELIGIBILITY:
Inclusion Criteria:

* Acute wounds in granulation phase with a minimum surface of 100cm2
* ≥ 18 years
* signing informed consent form
* guarantee adherence to protocol

Exclusion Criteria:

* chronic arterial insufficiency
* pregnant patients, lactating women or fertile adults that they don't use an effective contraceptive method
* involved in other assay
* previous disease; kidney, heart, hepatic, systemic or immune
* inability to understand informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
serious adverse events | 12 months
inflammatory changes | 12 months

SECONDARY OUTCOMES:
wound evaluation | 12 months
  inflammatory condition of the wound,surface,
immunological evaluation | 12 months
  anti Human Leukocyte Antigen 1 (HLA1),Short Tandem Repeat (STRS) detection
histological evaluation | 12 months
  Transforming growth factor beta 1 or Transforming growth factor beta (TGFB),wound biopsy
microbiological evaluation | 12 months
  microbiological culture

CONTACTS AND LOCATIONS:
Overall Officials: Gregorio Castellanos Escrig, MD, Principal Investigator — Hospital Clinico Universitario Virgen de la Arrixca
Locations (1):
- Gregorio Castellanos Escrig MD, Murcia, El Palmar, Spain